CLINICAL TRIAL: NCT00572975
Title: MALABSORPTION BLOOD TEST: Toward a Novel Approach to Quantify Steatorrhea
Brief Title: Malabsorption Blood Test:Toward a Novel Approach to Quantify Steatorrhea
Acronym: MBT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: Solvay Pharmaceuticals (Industry)
Responsible Party: Maria R. Mascarenhas, M.D., The Children's Hospital of Philadelphia
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2004-5-3733
Record Dates: First submitted 2007-12-11; First posted 2007-12-13 (Estimated); Last update posted 2008-09-30 (Estimated); Status verified 2008-09

CONDITIONS: Cystic Fibrosis; Pancreatic Insufficiency
Keywords: New diagnostic test for Cystic Fibrosis.
MeSH Terms: conditions — Cystic Fibrosis; Exocrine Pancreatic Insufficiency | interventions — pentadecanoic acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental)
  Interventions: Other: Pentadecanoic acid (PA) and Triheptadecanoin (THA)

INTERVENTIONS:
Other: Pentadecanoic acid (PA) and Triheptadecanoin (THA) — Two fats (Pentadecanoic acid and Triheptadecanoin) are administered in a breakfast shake for the purposes of determining malabsorption.
  in breakfast shake x1

SUMMARY:
*The purpose of this study is to develop a more accurate, reliable, specific and more acceptable alternative clinical test to the 72-hour stool and diet collection for quantifying fat malabsorption in people with CF and pancreatic insufficiency.

DETAILED DESCRIPTION:
* Nine subjects with CF will be recruited to complete the MBT on two separate occasions, with different doses of pancreatic enzymes
* At each MBT visit, subjects will receive a specific enzyme dose just before they drink the test meal (shake)
* Fat absorption is maximized when the enzymes are taken with the shake.
* If subjects usually receive brands of pancreatic enzymes different from Creon, their dose will be converted to an equivalent dose of Creon 20 for the study.

Prior to each study visit all subjects will be required to:

* Eat their usual diet for 2 days prior to MBT
* Refrain from consuming alcohol or dairy products for 24 hours prior to MBT
* Refrain from non-routine physical exercise for 20 hours prior to MBT
* Adhere to a 12-hour fast prior to MBT (from 8 PM previous night)
* Can drink water from 8:00 PM on the night before the test to 2:00 AM on the day of the test
* At visits 1 and 2, blood samples will be obtained at hourly intervals over a period of eight hours.
* Samples will be analyzed for PA, HA and Triglyceride concentrations.
* Patients will be permitted to ingest non-caloric and non-caffeinated beverages.
* At hour 6, patients will be provided 1000 Kcal, low fat (12 grams of fat) lunch meal.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with cystic fibrosis and pancreatic insufficiency (n=9), 8 years of age or older, in usual state of good health will be eligible to participate in this Aim.
* Subjects will be screened for genotype and a history of pancreatic insufficiency (PI). PI will be confirmed by measurement of fecal elastase 1< 200 mg/g stool.

Exclusion Criteria:

* Subjects will be ineligible if they have an FEV1 % predicted of < 40%, a history of fibrosing colonopathy or any significant bowel resection (>10 cm) with the exception of a routine, uncomplicated appendectomy.
* Subjects with diabetes mellitus or disorders associated with altered energy metabolism (i.e. hypothyroidism), or any major illnesses that affect the gastrointestinal tract, will not be eligible for the study.
* Subjects with significant liver disease, or significant developmental delay will also be excluded.
* Subjects will be excluded if they have a food allergy related to any components of the experimental shake (i.e., soy or chocolate) or the stool marker, carmine red.
* Subjects who are pregnant are not eligible. Subjects with a history of intolerance or allergy to Creon 20 will be excluded from the study.

Min Age: 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2006-08; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Aim 1:Comparing Gastric Emptying and Small Bowel Transit Protocol in Healthy Controls | 72 hours

SECONDARY OUTCOMES:
Aim 2:The results will establish which pattern of timing of enzyme ingestion results in optimal fat absorption of PA and HA. The results will also elucidate the role of gastric emptying and small bowel transit in subjects in CF. | 12-hour fast on 4 separate occasions, each at least 5 days apart
Aim 3: The results will establish the reproducibility of MBT as well as estimate the fecal loss of odd chain fatty acids (PA & THA) | 12-hour fast on three separate occasions, each at least 5 days apart
Aim 4: Dosage Titration Protocol is being tested in order to see changes in absorption with MBT | 12-hour fast on two separate occasions

CONTACTS AND LOCATIONS:
Overall Officials: Maria Mascarenhas, M.D., Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States